CLINICAL TRIAL: NCT02087579
Title: Open-Label Pharmacokinetic Study to Evaluate the Steady-State Venous and Capillary Plasma Concentrations of Five Antipsychotics: Aripiprazole, Olanzapine, Paliperidone, Quetiapine and Risperidone
Brief Title: Parallel Group, Multiple Dose Pharmacokinetics Study of Five Antipsychotic Medications in Psychiatric Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR103695; 2013-005289-20 (EudraCT Number); INDIGOAPS1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-02-17; First posted 2014-03-14 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Psychotic Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder
Keywords: Psychotic Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder; Antipsychotics; Aripiprazole; Olanzapine; Paliperidone; Quetiapine; Risperidone; Capillary Concentration
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder | interventions — Aripiprazole; Dosage Forms; Olanzapine; Paliperidone Palmitate; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort A: Aripiprazole (Experimental): Administration of oral formulation will continue at a participant's usual dose and dosing schedule.
  Interventions: Drug: Aripiprazole, oral formulation
- Cohort B: Olanzapine (Experimental): Administration of oral formulation will continue at a participant's usual dose and dosing schedule.
  Interventions: Drug: Olanzapine, oral formulation
- Cohort C: Paliperidone (Experimental): Administration of prolonged-release (extended-release) tablets or long-acting injectables (LAI) will continue at a participant's usual dose and dosing schedule.
  Interventions: Drug: Paliperidone, oral formulation; Drug: Paliperidone, LAI
- Cohort D: Quetiapine (Experimental): Administration of oral formulation will continue at a participant's usual dose and dosing schedule.
  Interventions: Drug: Quetiapine, oral formulation
- Cohort E: Risperidone (Experimental): Administration of oral formulation or LAI will continue at a participant's usual dose and dosing schedule.
  Interventions: Drug: Risperidone, oral formulation; Drug: Risperidone, LAI

INTERVENTIONS:
Drug: Aripiprazole, oral formulation — Aripiprazole tablets will be administered orally (by mouth), at no dose restriction, as per the locally approved label indications.
  Arms: Cohort A: Aripiprazole
Drug: Olanzapine, oral formulation — Olanzapine tablets will be administered orally, at no dose restriction as per the locally approved label indications.
  Arms: Cohort B: Olanzapine
Drug: Paliperidone, oral formulation — Paliperidone prolonged-release/extended-release (XR) formulation tablets will be administered orally, at no dose restriction, as per the locally approved label indications.
  Other Names: INVEGA®
  Arms: Cohort C: Paliperidone
Drug: Paliperidone, LAI — Paliperidone long-acting injectable (LAI) i.e., paliperidone palmitate injections, will be administered per the locally approved label indications.
  Other Names: INVEGA®
  Arms: Cohort C: Paliperidone
Drug: Quetiapine, oral formulation — Quetiapine immediate-release (IR) formulation or extended-release (XR) formulation tablets will be administered orally, at no dose restriction, as per the locally approved label indications.
  Arms: Cohort D: Quetiapine
Drug: Risperidone, oral formulation — Risperidone tablets will be administered orally, at no dose restriction, as per the locally approved label indications.
  Other Names: RISPERDAL®
  Arms: Cohort E: Risperidone
Drug: Risperidone, LAI — Risperidone LAI injections will be administered will be administered per the locally approved label indications.
  Other Names: RISPERDAL®
  Arms: Cohort E: Risperidone

SUMMARY:
The purpose of this study is to gather information about the steady-state plasma concentrations of aripiprazole, olanzapine, quetiapine and their relevant metabolites, at various dose levels and at different time points after dosing. In addition, comparison of capillary drug concentrations vs. venous drug concentrations will be performed for aripiprazole, olanzapine, paliperidone, quetiapine, risperidone and their relevant metabolites.

DETAILED DESCRIPTION:
This is an open-label (physicians and participants know the identity of the assigned treatment), parallel-group, multiple-dose, multicenter study to assess pharmacokinetics (what the body does to the medication) of five antipsychotics (APS) drugs: aripiprazole, olanzapine, paliperidone, quetiapine and risperidone in psychiatric participants who are receiving stable doses of these drugs for the treatment of their disease.

Pharmacokinetics data will be generated from venous and fingerstick-based capillary plasma concentrations of the drugs and their metabolites. The total number of enrolled participants in this study will be at least 265. Seventy-five participants will be enrolled for the aripiprazole, olanzapine and quetiapine cohorts (groups) each, and 20 participants will be enrolled for the paliperidone and risperidone cohorts each. In aripiprazole, olanzapine and quetiapine cohorts there will be two subgroups. Subgroup one, 20 participants for fingerstick capillary + venous blood sampling and subgroup two, 55 participants for only venous sampling. Paliperidone and risperidone cohorts will be subjected only to capillary + venous blood sampling.

The study will consist of a screening phase (within 21 days before Day 1) followed by a 3-day observation phase (Day 1 to Day 3). Participants will be admitted to the study center in the evening of Day -1 and will remain in the study center until discharged on Day 3 after completion of the last study-related procedure. During the observation phase, the administration of the prior antipsychotic medication will continue at a participant's usual dose and dosing schedule, under direct observation of the study staff. There will be no modification of the participant's medication during the study. Safety will be evaluated throughout the study and a mandatory pharmacogenomic blood sample will be collected for analysis of genes that may influence exposure of the APS studied.

ELIGIBILITY:
Inclusion Criteria:

* Must be clinically stable as per the investigator's judgment (no suicidal behavior or current significant suicidal judgment based on C-SSRS rating scale)
* No hospitalization for exacerbation of psychiatric symptoms during 3 months before screening
* Receiving treatment with aripiprazole, olanzapine, paliperidone, quetiapine or risperidone, or their combination before the study
* Must have body mass index between 17 and 40 kg/m2 (inclusive), and body weight not less than 47 kg
* Except for the indication for which the antipsychotic treatment is given, generally healthy with no clinically significant or unstable medical problems
* Must be able to give informed consent

Exclusion Criteria:

* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening as determined by the investigator
* Administering of strong inhibitors or inducers of CYP3A4, CYP2D6 enzymes, like fluoxetine
* History of or current clinically significant (particularly unstable) medical illness other than the indication
* Donated blood or blood products or had substantial loss of blood (more than 450 mL) within 3 months before Day -1
* Lack of 6 suitable puncture sites for capillary blood draws

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Aripiprazole concentration in venous and capillary plasma | 14 time points over 3 days postdose
  Venous blood samples will be collected at 8 scheduled time points after dosing and compared to fingerstick-based capillary blood samples collected at 6 scheduled time points after dosing.
Paliperidone concentration in venous and capillary plasma | 14 time points over 3 days postdose
Olanzapine concentration in venous and capillary plasma | 14 time points over 3 days postdose
Quetiapine concentration in venous and capillary plasma | 14 time points over 3 days postdose
Risperidone concentration in venous and capillary plasma | 14 time points over 3 days postdose

SECONDARY OUTCOMES:
Number of participants with an adverse event as a measure of safety | Participants will be followed for the duration of hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (24):
- United States (6):
  - Garden Grove, California
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Cedarhurst, New York
  - Austin, Texas
- Argentina (4):
  - Banfield
  - Buenos Aires
  - Córdoba
  - La Plata
- Belgium (4):
  - Aalst
  - Antwerp
  - Brussels
  - Kortenberg
- Brazil (2):
  - Rio de Janeiro
  - Valinhos
- Burgas, Bulgaria
- Germany (3):
  - Berlin
  - Hamburg
  - Lübeck
- Spain (4):
  - Badajoz
  - Barcelona
  - Torrevieja
  - Zamora

REFERENCES:
- See also: Open-Label Pharmacokinetic Study to Evaluate the Steady-State Venous and Capillary Plasma Concentrations of 5 Antipsychotics: Aripiprazole, Olanzapine, Paliperidone, Quetiapine and Risperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=6425&filename=CR103695_CSR.pdf